CLINICAL TRIAL: NCT01443910
Title: Weight Management Interactions in a Virtual Clinical Environment
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110238; 11-HG-0238
Record Dates: First submitted 2011-09-10; First posted 2011-09-30 (Estimated); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Healthy Volunteers; Body Weight
Keywords: Body Weight; Healthy Volunteer; Natural History
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- behavior, supportive: receiving information about behavior with supportive provider communication
- behaviors, directive: receiving information about behavior with directive provider communication
- genetics, directive: receiving information about genetics with directive provider communication
- genetics, supportive: receiving information about genetics with supportive provider communication

SUMMARY:
This study is part of an effort to learn about interactions between doctors and patients. We aim to understand how women feel about techniques that doctors use to talk with patients about their weight. We are studying women s reactions to these techniques using a virtual reality version of a doctor s office to create as realistic a model of a doctor s visit as possible. This can help us better understand what happens during real doctor s visits.

Women between the ages of 20 and 50 who are currently overweight may be eligible for this study. Participants will be recruited from the Washington D.C. area. This is not a weight treatment study.

Participants undergo the following procedures:

* Complete an online questionnaire about themselves, their experiences, and their thoughts about their weight
* Participate in activities in a virtual reality environment in which they interact with a virtual doctor in a virtual clinical scenario. For this experiment, participants wear a head-mounted display that allows them to see the virtual world images.
* Fill out a questionnaire after completing the virtual reality activities. This questionnaire includes information on the participants' virtual reality experience, the information provided in the experience, and additional questions about themselves and their thoughts.

DETAILED DESCRIPTION:
The primary goal of this research project is to build an evidence base related to primary care encounters that include discussions about a patient s body weight. We are particularly interested in how encounters impact patients health-related and weight-related attitudes and beliefs. Furthermore, this project aims to determine how a physician s approach to the health care encounter impacts its outcome.

The current study is a controlled experiment in which participants will be participate in a weight counseling encounter with a virtual reality-based doctor. The virtual doctor will present weight etiology information. Participants will fill out a self-report questionnaire online, prior to this encounter. They will then come in to the Immersive Virtual Environment Testing Area in the NIH Clinical Center for a visit. During this visit, they will engage in the interaction with the virtual doctor and then fill out a post-test questionnaire. Participants in the main trial will include approximately 222 healthy adult females between 20-50 years of age who have a BMI of greater than or equal to 25 and are dissatisfied with their current weight.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. being between 20 and 50 years old
  2. having a self-reported body mass index of greater than or equal to 25
  3. having the ability to read, write, and converse in English
  4. being able to come to the NIH Clinical Center for one visit

EXCLUSION CRITERIA:

1. having a vestibular or seizure disorder
2. having a high propensity for motion sickness
3. known pregnancy
4. uncorrected low vision or hearing
5. inability to complete tasks in the virtual environment
6. being an NHGRI employee
7. being or training to become a health care provider

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Overweight, adult women will participate in a weight counseling encounter with a virtual reality-based doctor
Sampling Method: Non-Probability Sample
Enrollment: 318 (Actual)
Dates: Start 2012-02-29 (Actual); Primary Completion 2016-04-06 (Actual); Study Completion 2016-04-06 (Actual)

PRIMARY OUTCOMES:
attitudes, beliefs, and behavior | cross-sectional
  self-report outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Susan Persky, Ph.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Agurs-Collins T, Khoury MJ, Simon-Morton D, Olster DH, Harris JR, Milner JA. Public health genomics: translating obesity genomics research into population health benefits. Obesity (Silver Spring). 2008 Dec;16 Suppl 3(Suppl 3):S85-94. doi: 10.1038/oby.2008.517. PMID 19037221
- [Background] Kumanyika SK, Van Horn L, Bowen D, Perri MG, Rolls BJ, Czajkowski SM, Schron E. Maintenance of dietary behavior change. Health Psychol. 2000 Jan;19(1S):42-56. doi: 10.1037/0278-6133.19.suppl1.42. PMID 10709947
- [Background] Kushner RF. Understanding obesity by asking the right questions. Perspect Biol Med. 2010 Winter;53(1):148-51. doi: 10.1353/pbm.0.0139. PMID 20201162
- [Derived] Persky S, Street RL Jr. Evaluating Approaches for Communication About Genomic Influences on Body Weight. Ann Behav Med. 2015 Oct;49(5):675-84. doi: 10.1007/s12160-015-9701-8. PMID 25894275
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-HG-0238.html